CLINICAL TRIAL: NCT05038397
Title: A Study to Evaluate Efficacy and Safety of TheraSphere and Resection Combination Therapy in Patients With Single Large ((> 5 cm, Long Diameter ) Hepatocellular Carcinoma : Exploratory Trial
Brief Title: A Study to Evaluate Efficacy and Safety of TheraSphere and Resection Combination Therapy in Patients With Single Large ((> 5cm, Long Diameter ) Hepatocellular Carcinoma : Exploratory Trial
Acronym: Therasphere
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedicalExcellence (Other)
Collaborators: BTG International Inc. (Other); Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTG-SP-21.028-F01
Record Dates: First submitted 2021-08-13; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therasphere (Experimental)
  Interventions: Device: Theraspere

INTERVENTIONS:
Device: Theraspere — Prior to the administration of TheraSphere, the patient should undergo hepatic arterial catheterization using balloon catheterization or other appropriate angiographic techniques to prevent extrahepatic shunting. Following the placement of the hepatic catheter, 75 MBq to 150 MBq (2 mCi to 4 mCi) of Tc-99m MAA is administered into the hepatic artery to determine the extent of A-V shunting to the lungs and to confirm the absence of gastric and duodenal flow. When the possibility of extrahepatic shunting has been evaluated and the patient deemed acceptable for treatment, TheraSphere may be administered.

SUMMARY:
A study to evaluate efficacy and safety of TheraSphere and resection combination therapy in patients with single large ((> 5cm, long diameter ) hepatocellular carcinoma :

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the sixth most common cancer and the third leading cause of cancer related death worldwide. Because HCC usually occurs in patients with underlying liver disease, candidates for treatment strategies should be selected based on tumor status and liver function. According to the Barcelona Clinic Liver Cancer (BCLC) staging system, which is widely used for treatment allocation , hepatic resection is considered the treatment of choice for single tumors without macrovascular invasion or extrahepatic spread. These patients are beyond the Milan criteria; liver transplantation is not recommended as the first treatment choice because of the risk of recurrence and the scarcity of donors. Ablative therapies, such as percutaneous ethanol injection and radiofrequency ablation (RFA), rarely achieve complete necrosis in tumors > 3 cm.

Consequently, hepatic resection is considered the only po tentially curative treatment for these patients. Nevertheless, few patients are candidates for hepatic resection because of associated liver cirrhosis and the risk of inducing postoperative liver decompensation. Although perioperative mortality of hepatic resection in cirrhotic patients has decreased, candidates must be selected carefully to avoid life threatening complications. The lon g term outcome of hepatic resection remains poor, mainly because tumors often recur after resection. Moreove r, s ingle large ( 5cm) tumor showed significantly worse survival than other BCLC stage A, which indicate that single tumor should be differently staged according to their tumor size . For these reasons, whether hepatic resection is the optimal treatment for large single HCCs is a matter of debate.

Yttrium 9 0 radioembolization (Y90) allow s accurate tumor targeting while spa ring surrounding parenchyma, resulting in down staging potential and bridging to transplantation strategies The responsiveness of HCC to radiation, while long recognized, has been limited by nontargeted tissue exposure and radiation injury. With the devel opment of advanced microcatheters and short radius of emission of Y90, single lesions confined to particular liver segment s may now be approached with s uperselective radiotherapy, permitting ablative doses to a confined liver volume. The purpose of this study i s to assess the efficacy and safety of neo adjuvant Therapsphere to down stage in single large ( (> 5cm , long diameter HCC treated with resection.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Clinical or histological diagnosis of HCC based on the guidelines of the American Association for the Study of Liver Diseases (AASLD).
3. Single large (> 5cm, long diameter) lesion that is typically enhanced* and bi-dimensionally measurable by multiphasic spiral CT scan and dynamic contrast-enhanced MRI.
4. Tumor conditions confirmed by abdominal imaging (contrast enhanced CT ± MRI) performed within 28 days prior to the enrollment
5. Age of at least 19 years.
6. ECOG Performance Status of 0.
7. Child-Pugh class A (Child-Pugh score ≤6).
8. Life expectancy of at least 16 weeks.
9. Patients with bile duct involvement can be enrolled if patients have adequate bone marrow, liver, and renal function
10. Adequate bone marrow, liver as assessed by the following laboratory requirements (no transfusion, no restoration), conducted screening: Data can be used within 28 days of screening.

    * Hemoglobin ≥ 8.0g/dL
    * Absolute neutrophil count (ANC) ≥ 1,000/mm3
    * Platelet count ≥ 100,000/μL
    * Total bilirubin ≤ 2mg/dL
    * Serum albumin ≥ 3g/dL
    * ALT and AST < 5 × upper limit of normal
    * PT-INR ≤ 1.7
11. Patients with involvement with tumor thrombus in the second-order branches of the portal vein or distal to the second-order branches (Vp1-Vp2) can be enrolled if operability is confirmed by the surgeon.

Exclusion Criteria:

1. Diffuse infiltrative tumor type
2. Presence of separate daughter nodule
3. Poorly defined and/or mixed-irregular tumor margin
4. Definitive combined HCC-cholangiocarcinoma on images
5. A history of receiving any systemic therapy of the molecularly targeted agents, immunotherapy, external beam radiation to the liver or cytotoxic chemotherapy for the treatment of HCC
6. Presence of extrahepatic HCC: Involvement of vessels [major branch of hepatic vein invasion; major branch of portal vein invasion from the first order portal vein branch (Vp3) to main portal vein (Vp4)]; lymph node, metastasis
7. History or presence of hepatic encephalopathy
8. Ascites, moderate, large or intractable
9. Active clinically serious infections (> grade 2, NCI-CTCAE version 4.02), including spontaneous bacterial peritonitis.
10. Untreated active chronic hepatitis B
11. Esophageal or gastric varices ≥ F2 (grade 2) with red color sign positive without prophylaxis (non-selective beta-blocker or endoscopic variceal ligation) or history of variceal bleeding without endoscopic variceal ligation/ injection sclerosis
12. Active ulcer of stomach or duodenum: untreated or presence of visible vessel
13. Any major surgery within 4 weeks, or any minor surgery within 2 weeks prior to signing the informed consent form
14. Candidate for liver transplantation and/or a history of liver transplantation
15. History of cardiac diseases: congestive heart failure greater than NYHA class 2; active coronary artery disease (myocardial infarction more than 6 months prior to study entry is allowed); uncontrolled hypertension and diabetes mellitus
16. History of AIDS/HIV infection
17. Seizure disorder requiring medication (such as steroids or anti-epileptics)
18. History of organ allograft
19. Evidence or history of bleeding diathesis, or thromboembolic events requiring treatment
20. Current renal dialysis
21. Previous or concurrent cancer that has a primary site or histology distinct from HCC, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis, and T1] or any cancer curatively treated less than 3 years prior to enrollment.
22. (Deleted)
23. Tc-99m macroaggregated albumin (MAA) hepatic arterial perfusion scintigraphy shows any deposition to the gastrointestinal tract that may not be corrected by angiographic techniques.
24. Shunting of blood to the lungs that could result in delivery of greater than 16.5 mCi of yttrium-90 to the lungs. Radiation pneumonitis has been seen in patients receiving doses to the lungs greater than 30 Gy in a single treatment.
25. Hepatic artery catheterization is contraindicated; such as patients with vascular abnormalities or bleeding diathesis.
26. Severe liver dysfunction or pulmonary insufficiency
27. Pregnant or breast feeding women, or impossible to use of reliable methods of contraception
28. Subject who the investigator deems inappropriate to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) after resection | 96 Weeks

SECONDARY OUTCOMES:
Overall survival (OS) after resection | 96 Weeks
Time to recurrence (TTR) of tumor after resection : | 96 Weeks
Safety profiles | 96 Weeks
  Frequency of Adverse events
Rate of post operative hepatic decompensation | 96 Weeks
  Hepatic decompensation was defined as incidence of both jaundice (serum bilirubin ≥ 5 mg/dL) and coagulopathy (prothrombin time < 40%) with or without the presence of ascites and/or encephalopathy as determined at physical examination [Hepatol Int 2009;3(1):269-282].

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea